CLINICAL TRIAL: NCT06737614
Title: Can Pulse Pressure Assessment at the Bedside Detect Low Values or Track Changes of Stroke Volume in Critically Ill Patients? The Multicenter, Cross-sectional, Observational, ANDROMEDA-PEGASUS Study
Brief Title: Relationship Between Pulse Pressure and Stroke Volume in the Critically Ill Patients: The ANDROMEDA-PEGASUS Study
Status: Recruiting | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Erasmus Medical Center (Other); Fundacion Clinica Valle del Lili (Other); Hospital do Coracao (Other)
Responsible Party: Sponsor
Other Study IDs: 240730006
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2024-12

CONDITIONS: Critical Illness
Keywords: pulse pressure; stroke volume
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this study is to assess the predictive capacity of pulse pressure to estimate stroke volume, as assessed by bedside echocardiography in critically ill patients.

We hypothesize that pulse pressure will be able to adequately detect low values of stroke volume, and to track changes of stroke volume during commonly used dynamic cardiovascular interventions.

Pulse pressure transduced from an arterial line will be measured simultaneously with left ventricular outflow tract velocity time integral in a broad range of critically ill patients. Ancillary clinical, hemodynamic and echocardiographic data will also be registered.

DETAILED DESCRIPTION:
Critically ill patients often present complex cardiovascular derangements that impair oxygen delivery to the tissues leading to progressive organ dysfunction. Monitoring tissue perfusion and identifying the predominant hemodynamic patterns are key clinical objectives to implement resuscitative strategies and revert this vicious cycle. However, in different stages of acute circulatory dysfunction at the emergency department (ED) or the intensive care unit (ICU), or resource-limited settings, initial resuscitative decisions may be taken with basic clinical information only. In addition, many therapeutic interventions in the ICU such as fluids, diuretics, vasoactive drugs, and ventilatory-related maneuvers, among others, may jeopardize stroke volume (SV) in different ways, a fact that may evolve undetected due to the absence of specific hemodynamic monitors in all patients.

Unfortunately, there is no simple, costless, and universally available clinical monitor to detect low SV. There have been, however, physiological implications to use blood pressure components as a surrogate for SV. Although pulse pressure (PP) has been observed to be largely determined by SV in experimental conditions, the key issues remain to be clarified: can PP monitoring at the bedside be useful to detect extreme values, or track changes, in underlying SV? Moreover, what are the limitations, the contexts, the technical aspects, among other factors, that can affect this relationship, and thus help clinicians to potentially use PP as an early warning signal or a trigger for initial resuscitative or therapeutic interventions?

From a clinical point of view, the most relevant question is if PP monitoring can detect a low SV so that corrective measures might be implemented, while more advanced confirmatory monitoring, including point-of-care ultrasound, is pending. In addition, what are the potential confounders for this assumption? If these questions are answered, this simple and costless tool may be used as a first-line approach for macrohemodynamic profiling and clinical decision-making, which could be especially valuable in resource-limited settings and in sites where ultrasound or advanced cardiac output monitoring is not immediately available. In this multicenter, observational, cross-sectional study, we aim at answering the following research question:

Research Question

* In critically ill patients, does pulse pressure, measured through an invasive arterial line, have an adequate predictive capacity to estimate stroke volume, as assessed by bedside echocardiography?
* We hypothesize that pulse pressure will be able to adequately detect low values of stroke volume, and to track changes of stroke volume during commonly used dynamic cardiovascular interventions.

Primary Objective

- To assess the predictive capacity of pulse pressure to detect low stroke volume, evaluated by bedside ultrasonography in critically ill patients.

Secondary Objectives

* To assess the predictive capacity of PP to detect low SV in different clinical contexts in ICU patients, such as in those with acute respiratory distress syndrome (ARDS), postoperative states, or septic shock, among others.
* To assess the impact of several demographic, clinical and technical issues on the predictive capacity of PP to estimate SV, such as mechanical ventilation, vasoactive medication, age, position of the arterial line, among others.
* To determine the capacity of PP to track changes of SV during common intensive care interventions such as passive leg raising (PLR) maneuver or fluid challenges.

ELIGIBILITY:
Inclusion Criteria:

* 18 years
* Admitted to ICU
* Functioning arterial line in place

Exclusion Criteria:

* Pregnancy
* Inadequate arterial line transduction (see below)
* Refusal of consent
* Patient who requires extracorporeal circulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - During the study period (one or two weeks according to local study team), eligible patients will be identified during morning rounds. Consecutive patients which comply with inclusion and exclusion criteria and consent in participating will be included in the study. A broad range of ICU patients will be included to perform relevant subgroup analysis.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Left ventricular outflow tract velocity time integral | 1 day
  measured by bedside echocardiography
Pulse pressure | 1 day
  measured from invasive arterial line

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Kattan, MD, PhD, Principal Investigator — Assistant Professor; Glenn Hernandez, MD, PhD, Principal Investigator — Full Professor
Locations (3):
- Hospital Do Coracao, São Paulo, Brazil
- Hospital Clinico UC Christus, Santiago, Chile
- Fundacion Valle del Lili, Cali, Colombia

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared upon reasonable request to the principal investigators
Supporting Information: Study Protocol, SAP
Time Frame: after publication
Access Criteria: De-identified data may be shared upon reasonable request to the principal investigators

REFERENCES:
- [Background] Bakker J, Kattan E, Annane D, Castro R, Cecconi M, De Backer D, Dubin A, Evans L, Gong MN, Hamzaoui O, Ince C, Levy B, Monnet X, Ospina Tascon GA, Ostermann M, Pinsky MR, Russell JA, Saugel B, Scheeren TWL, Teboul JL, Vieillard Baron A, Vincent JL, Zampieri FG, Hernandez G. Current practice and evolving concepts in septic shock resuscitation. Intensive Care Med. 2022 Feb;48(2):148-163. doi: 10.1007/s00134-021-06595-9. Epub 2021 Dec 15. PMID 34910228
- [Background] Hernandez G, Ospina-Tascon GA, Damiani LP, Estenssoro E, Dubin A, Hurtado J, Friedman G, Castro R, Alegria L, Teboul JL, Cecconi M, Ferri G, Jibaja M, Pairumani R, Fernandez P, Barahona D, Granda-Luna V, Cavalcanti AB, Bakker J; The ANDROMEDA SHOCK Investigators and the Latin America Intensive Care Network (LIVEN); Hernandez G, Ospina-Tascon G, Petri Damiani L, Estenssoro E, Dubin A, Hurtado J, Friedman G, Castro R, Alegria L, Teboul JL, Cecconi M, Cecconi M, Ferri G, Jibaja M, Pairumani R, Fernandez P, Barahona D, Cavalcanti AB, Bakker J, Hernandez G, Alegria L, Ferri G, Rodriguez N, Holger P, Soto N, Pozo M, Bakker J, Cook D, Vincent JL, Rhodes A, Kavanagh BP, Dellinger P, Rietdijk W, Carpio D, Pavez N, Henriquez E, Bravo S, Valenzuela ED, Vera M, Dreyse J, Oviedo V, Cid MA, Larroulet M, Petruska E, Sarabia C, Gallardo D, Sanchez JE, Gonzalez H, Arancibia JM, Munoz A, Ramirez G, Aravena F, Aquevedo A, Zambrano F, Bozinovic M, Valle F, Ramirez M, Rossel V, Munoz P, Ceballos C, Esveile C, Carmona C, Candia E, Mendoza D, Sanchez A, Ponce D, Ponce D, Lastra J, Nahuelpan B, Fasce F, Luengo C, Medel N, Cortes C, Campassi L, Rubatto P, Horna N, Furche M, Pendino JC, Bettini L, Lovesio C, Gonzalez MC, Rodruguez J, Canales H, Caminos F, Galletti C, Minoldo E, Aramburu MJ, Olmos D, Nin N, Tenzi J, Quiroga C, Lacuesta P, Gaudin A, Pais R, Silvestre A, Olivera G, Rieppi G, Berrutti D, Ochoa M, Cobos P, Vintimilla F, Ramirez V, Tobar M, Garcia F, Picoita F, Remache N, Granda V, Paredes F, Barzallo E, Garces P, Guerrero F, Salazar S, Torres G, Tana C, Calahorrano J, Solis F, Torres P, Herrera L, Ornes A, Perez V, Delgado G, Lopez A, Espinosa E, Moreira J, Salcedo B, Villacres I, Suing J, Lopez M, Gomez L, Toctaquiza G, Cadena Zapata M, Orazabal MA, Pardo Espejo R, Jimenez J, Calderon A, Paredes G, Barberan JL, Moya T, Atehortua H, Sabogal R, Ortiz G, Lara A, Sanchez F, Hernan Portilla A, Davila H, Mora JA, Calderon LE, Alvarez I, Escobar E, Bejarano A, Bustamante LA, Aldana JL. Effect of a Resuscitation Strategy Targeting Peripheral Perfusion Status vs Serum Lactate Levels on 28-Day Mortality Among Patients With Septic Shock: The ANDROMEDA-SHOCK Randomized Clinical Trial. JAMA. 2019 Feb 19;321(7):654-664. doi: 10.1001/jama.2019.0071. PMID 30772908
- [Background] Hernandez G, Messina A, Kattan E. Invasive arterial pressure monitoring: much more than mean arterial pressure! Intensive Care Med. 2022 Oct;48(10):1495-1497. doi: 10.1007/s00134-022-06798-8. Epub 2022 Jul 8. No abstract available. PMID 35802139
- [Background] Westerhof N, Lankhaar JW, Westerhof BE. The arterial Windkessel. Med Biol Eng Comput. 2009 Feb;47(2):131-41. doi: 10.1007/s11517-008-0359-2. Epub 2008 Jun 10. PMID 18543011
- [Background] Marquez J, McCurry K, Severyn DA, Pinsky MR. Ability of pulse power, esophageal Doppler, and arterial pulse pressure to estimate rapid changes in stroke volume in humans. Crit Care Med. 2008 Nov;36(11):3001-7. doi: 10.1097/CCM.0b013e31818b31f0. PMID 18824912
- [Background] Convertino VA, Cooke WH, Holcomb JB. Arterial pulse pressure and its association with reduced stroke volume during progressive central hypovolemia. J Trauma. 2006 Sep;61(3):629-34. doi: 10.1097/01.ta.0000196663.34175.33. PMID 16966999